CLINICAL TRIAL: NCT05101096
Title: A Phase 1/2 Open-Label Study of Sacituzumab Govitecan in Japanese Patients With Advanced Solid Tumors (ASCENT-J02)
Brief Title: Study of Sacituzumab Govitecan (SG) in Japanese Participants With Advanced Solid Tumors
Acronym: ASCENT-J02
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-569-6172; jRCT2031210346 (Registry Identifier: Japan Registry of Clinical Trials)
Record Dates: First submitted 2021-10-19; First posted 2021-11-01 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Advanced Solid Tumor; Metastatic Triple-Negative Breast Cancer; HR+/HER2- Metastatic Breast Cancer; Metastatic Urothelial Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — sacituzumab govitecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (8):
- Sacituzumab Govitecan-hziy 6 mg, Advanced Solid Tumors (Experimental): (Phase 1 Cohort A: dose escalation) Japanese participants with advanced solid tumors will receive sacituzumab govitecan-hziy (SG) 6 mg/kg by intravenous (IV) injection on Day 1 and Day 8 of a 21-day cycle until disease progression or unacceptable toxicity.
  Interventions: Drug: Sacituzumab Govitecan-hziy
- Sacituzumab Govitecan-hziy 8 mg, Advanced Solid Tumors (Experimental): (Phase 1 Cohort A: dose escalation) Japanese participants with advanced solid tumors will receive SG 8 mg/kg by IV injection on Day 1 and Day 8 of a 21-day cycle until disease progression or unacceptable toxicity.
  Interventions: Drug: Sacituzumab Govitecan-hziy
- Sacituzumab Govitecan-hziy 10 mg, Advanced Solid Tumors (Experimental): (Phase 1 Cohort A: dose escalation) Japanese participants with advanced solid tumors will receive SG 10 mg/kg by IV injection on Day 1 and Day 8 of a 21-day cycle until disease progression or unacceptable toxicity.
  Interventions: Drug: Sacituzumab Govitecan-hziy
- Sacituzumab Govitecan-hziy 6 mg, UGT1A1 Polymorphism (Experimental): (Phase 1 Cohort B: dose escalation) Japanese participants with UGT1A1 polymorphism will receive SG 6 mg/kg by IV injection on Day 1 and Day 8 of a 21-day cycle until disease progression or unacceptable toxicity.
  Interventions: Drug: Sacituzumab Govitecan-hziy
- Sacituzumab Govitecan-hziy 10 mg, UGT1A1 Polymorphism (Experimental): (Phase 1 Cohort B: dose escalation) Japanese participants with UGT1A1 polymorphism will receive SG 10 mg/kg by IV injection on Day 1 and Day 8 of a 21-day cycle until disease progression or unacceptable toxicity.
  Interventions: Drug: Sacituzumab Govitecan-hziy
- Sacituzumab Govitecan-hziy, Metastatic Triple-negative Breast Cancer (mTNBC) (Experimental): (Phase 2: dose expansion) Japanese participants with mTNBC will receive SG at the recommended Phase 2 dose (RP2D) on Day 1 and Day 8 of a 21-day cycle until disease progression or unacceptable toxicity.
  Interventions: Drug: Sacituzumab Govitecan-hziy
- Sacituzumab Govitecan-hziy, HR+/HER2- Metastatic Breast Cancer (HR+/HER2- mBC) (Experimental): (Phase 2) Japanese participants with HR+/HER2- mBC will receive SG at the recommended Phase 2 dose (RP2D) on Day 1 and Day 8 of a 21 day cycle until disease progression or unacceptable toxicity.
  Interventions: Drug: Sacituzumab Govitecan-hziy
- Sacituzumab Govitecan-hziy, Metastatic Urothelial Carcinoma (mUC) (Experimental): (Phase 2) Japanese participants with mUC will receive SG at the recommended Phase 2 dose (RP2D) on Day 1 and Day 8 of a 21 day cycle until disease progression or unacceptable toxicity.
  Interventions: Drug: Sacituzumab Govitecan-hziy

INTERVENTIONS:
Drug: Sacituzumab Govitecan-hziy — Administered intravenously (IV)
  Other Names: IMMU-132; Trodelvy™; GS-0132

SUMMARY:
The primary objectives of this study are as follows:

Phase 1 (sequential dose-escalation): to evaluate the safety and tolerability of sacituzumab govitecan-hziy (SG) as a single agent and to determine the recommended Phase 2 dose (RP2D) of SG in Japanese participants with advance solid tumors.

Phase 2: Evaluate the safety and efficacy of SG in Japanese participants with metastatic triple-negative breast cancer (mTNBC), hormone receptor-positive (HR+)/human epidermal growth factor receptor 2-negative (HER2-) metastatic breast cancer (mBC), and metastatic urothelial cancer (mUC).

ELIGIBILITY:
Key Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1
* Measurable disease by computed tomography (CT) or magnetic resonance imaging (MRI) as per RECIST Version 1.1 criteria
* Adequate hematologic counts without transfusional or growth factor support within 2 weeks of study drug initiation
* Adequate hepatic function (bilirubin ≤ 1.5 upper limit of normal (ULN)), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 ULN
* Creatinine clearance ≥ 30 mL/min
* Male and female individuals of childbearing potential who engage in heterosexual intercourse must agree to use protocol-specified method(s) of contraception.
* Phase 1 only: Histologically or cytologically confirmed advanced solid tumor that is refractory to or intolerant of all standard therapy or for which no standard therapy is available.
* Phase 2 metastatic triple-negative breast cancer (mTNBC) Cohort: Histologically or cytologically confirmed TNBC per American Society of Clinical Oncologists/College of American Pathologists (ASCO/CAP) criteria, based on the most recent analyzed biopsy or other pathology specimen. Refractory to or relapsed after at least 2 prior standard-of-care chemotherapy regimens for unresectable, locally advanced or metastatic breast cancer.
* Phase 2 hormone receptor-positive/human epidermal growth factor receptor 2-negative metastatic breast cancer (HR+/HER2- mBC) Cohort: Documented evidence of HR+/HER2- mBC confirmed by a local laboratory and defined per ASCO/CAP criteria.

  * Refractory to or relapsed after 2 prior systemic chemotherapy regimens for locally advanced unresectable or metastatic disease.
* Phase 2 metastatic urothelial cancer (mUC) Cohort: Histologically documented UC that is metastatic or locally advanced unresectable.

  * Progressed or recurred following receipt of platinum-containing regimen and anti-PD-1/PD-L1 therapy for metastatic or locally advanced unresectable disease

Key Exclusion Criteria:

* Positive serum pregnancy test, or females who may possibly be pregnant
* Known Gilbert's disease
* Have previously received antibody drug conjugate containing topoisomerase I inhibitors
* Presence of bulky disease (defined as any single mass > 7 cm in greatest dimension).
* Known to be HIV positive, or hepatitis B virus (HBV) surface antigen positive or hepatitis C virus (HCV) antibody positive at screening
* Known history of significant cardiac disease
* Known history of clinically significant active chronic obstructive pulmonary disease, or other moderate-to-severe chronic respiratory illness
* History of interstitial lung disease
* History of clinically significant gastrointestinal (GI) bleeding, have active chronic inflammatory bowel disease (ulcerative colitis, Crohn's disease) or GI perforation
* Individuals with a history of anaphylactic reaction to irinotecan.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2021-10-20 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Percentage of Participants Experiencing Treatment-emergent Adverse Events (TEAEs) Defined by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 4.03 | First dose date to last dose date (Up to 15 weeks) plus 30 days
Phase 1: Percentage of Participants Experiencing Laboratory Abnormalities Defined by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 4.03 | First dose date to last dose date (Up to 15 weeks) plus 30 days
Phase 1: Percentage of Participants Experiencing Dose-limiting toxicity (DLTs) per Dose level | First dose date up to 21 days
Phase 2:(Metastatic Triple-negative Breast Cancer (mTNBC);Hormone Receptor-positive/Human Epidermal Growth Factor Receptor 2-negative Metastatic Breast Cancer (HR+/HER2- mBC) Cohorts):Objective Response Rate (ORR) as Assessed by IRC | Up to 17 months
  ORR is defined as the proportion of participants who achieve a complete response (CR) or partial response (PR), confirmed at least 4 weeks later as assessed by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) as assessed by Independent Review Committee (IRC).
Phase 2 (Metastatic Urothelial Cancer (mUC) Cohort): ORR as Assessed by Investigator | Up to 17 months
  ORR is defined as the proportion of participants who achieve a complete response (CR) or partial response (PR) confirmed at least 4 weeks later as assessed by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)

SECONDARY OUTCOMES:
Phase 1: Pharmacokinetic (PK) Parameter: Cmax of Sacituzumab Govitecan-hziy (SG) and Free SN-38 | Up to 33 months
  Cmax is defined as the maximum observed concentration of drug
Phase 1: PK Parameter: Tmax of SG and Free SN-38 | Up to 33 months
  Tmax is defined as time (observed time point) of Cmax
Phase 1: PK Parameter: AUC0-168h of SG and Free SN-38 | Up to 33 months
  AUC0-168h is defined as partial area under the concentration of drug over time between 0 to time 168-hour.
Phase 1 : Percentage of Participants Who Develop Anti-Drug Antibodies (ADAs) Against SG | Up to 33 months
Phase 2 (All Cohorts): Percentage of Participants Experiencing TEAEs Defined by NCI CTCAE Version 4.03 | First dose date to last dose date (Up to 33 months) plus 30 days
Phase 2 (All Cohorts): Percentage of Participants Experiencing Laboratory Abnormalities Defined by NCI CTCAE Version 4.03 | First dose date to last dose date (Up to 33 months) plus 30 days
Phase 2(All Cohorts): Progression-free survival (PFS) as Assessed by Investigator | Up to 33 months
  PFS is defined as the interval from the first dose of SG to the earlier of the first documentation of objective progressive disease (PD) or death from any cause, whichever comes first.
Phase 2 (All Cohorts): ORR as Assessed by Investigator | Up to 17 months
  ORR is defined as the proportion of participants who achieve a CR or PR as assessed by RECIST v1.1.
Phase 2 (All Cohorts): Overall Survival (OS) | Up to 33 months
  OS is defined as the time from date of first dose of SG to death from any cause, whichever comes first.
Phase 2 (All Cohorts): Duration of Response (DOR) as Assessed by Investigator | Up to 33 months
  DOR is defined as the time from the first documentation of CR or PR to the earlier of the first documentation of objective PD or death from any cause.
Phase 2 (All Cohorts): Time to response (TTR) as Assessed by Investigator | Up to 17 months
  TTR is defined as the time from first dose of SG to the first documentation of CR or PR.
Phase 2 (mTNBC and HR+/HER2- mBC Cohorts): Progression-free survival (PFS) as Assessed by IRC | Up to 33 months
  PFS is defined as the interval from the first dose of SG to the earlier of the first documentation of objective progressive disease (PD) or death from any cause, whichever comes first.
Phase 2 (mTNBC and HR+/HER2- mBC Cohorts): Duration of Response (DOR) as Assessed by IRC | Up to 33 months
  DOR is defined as the time from the first documentation of CR or PR to the earlier of the first documentation of objective PD or death from any cause.
Phase 2 (mTNBC and HR+/HER2- mBC Cohorts): Time to response (TTR) as Assessed by IRC | Up to 17 months
  TTR is defined as the time from first dose of SG to the first documentation of CR or PR.

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (36):
- Japan (36):
  - Aichi Cancer Center Hospital, Aichi
  - Akita University Hospital, Akita
  - Tohoku University Hospital, Aoba-ku
  - Hirosaki University Hospital, Aomori
  - Kanagawa Cancer Center, Asahi-ku
  - Juntendo University Hospital, Bunkyō City
  - Chiba Cancer Center, Chiba
  - National Cancer Center Hospital East, Chiba
  - Chiba Cancer, Chūōku
  - Nagoya University Hospital, Chūōku
  - Osaka International Cancer Institute, Chūōku
  - Shikoku Cancer Center, Ehime
  - National Hospital Organization Shikoku Cancer Center, Ehime
  - Hyogo Cancer Center, Hyōgo
  - Kagawa University Hospital, Kagawa
  - Tokai University School of Medicine, Kanagawa
  - The Cancer Institute Hospital of JFCR, Kōtō City
  - Kumamoto University Hospital, Kumamoto
  - Kyoto University Hospital, Kyoto
  - Hiroshima University Hospital, Minamiku
  - Nara Medical University Hospital, Nara
  - Hyogo College of Medicine College Hospital, Nishinomiya-shi
  - Okayama University Hospital, Okayama
  - Osaka International Cancer Institute, Osaka
  - Osaka Metropolitan University Hospital, Osaka
  - Osaka University Hospital, Osaka
  - Kindai University Hospital, Osaka
  - Kindai University Hospital, Osakasayama-shi
  - Saitama Medical University, Saitama
  - National Hospital Organization Hokkaido Cancer Center, Sapporo
  - National Center for Global Health and Medicine, Shinjuku-ku
  - National Cancer Center hospital, Tokyo
  - Tokyo Medical And Dental University, Medical Hospital, Tokyo
  - Showa University Hospital, Tokyo
  - Keio University Hospital, Tokyo
  - Yamaguchi University Hospital, Yamaguchi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Naito Y, Nakamura S, Kawaguchi-Sakita N, Ishida T, Nakayama T, Yamamoto Y, Masuda N, Matsumoto K, Kogawa T, Sudo K, Shimomura A, Lai C, Zhang D, Iwahori Y, Gary D, Huynh D, Iwata H. Preliminary results from ASCENT-J02: a phase 1/2 study of sacituzumab govitecan in Japanese patients with advanced solid tumors. Int J Clin Oncol. 2024 Nov;29(11):1684-1695. doi: 10.1007/s10147-024-02589-x. Epub 2024 Sep 20. PMID 39302614
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=GS-US-569-6172